CLINICAL TRIAL: NCT04626271
Title: Evaluation of the Accuracy and Usability of the ACR | U.S. Urine Analysis Test System in the Lay User Hands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Healthy.io Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ACR-US-MCU-01
Record Dates: First submitted 2020-10-25; First posted 2020-11-12 (Actual); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Albuminuria
MeSH Terms: conditions — Albuminuria

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ACR | U.S. Urine Analysis Test System (Experimental): Urine samples are collected and tested by a lay user, using the new home use device. The lay user test results are compared to the results obtained by testing the same urine sample on the comparison device.
  Interventions: Device: ACR | U.S. Urine Analysis Test System; Device: URiSCAN Optima Urine Analyzer

INTERVENTIONS:
Device: ACR | U.S. Urine Analysis Test System — Each study participant will test their urine sample using the ACR | U.S. test device - a home-use device intended for the semi-quantitative measurement of ACR in the urine (albumin and creatinine ratio) and used to aid in the management of kidney health.
Device: URiSCAN Optima Urine Analyzer — Upon completion of the test using the ACR | U.S. device, each urine sample will be provided to a professional user for further urine analysis test using the comparator device, the URiSCAN Optima Urine Analyzer.

SUMMARY:
Eligible subjects meeting the pathological profile will be recruited at the designated site by the study personnel. Following subject consent, the subjects will be evaluated for eligibility based on their health condition and history.

The ACR | U.S. kit, in its original packaging, along with the ACR | U.S. smartphone application will be provided to the subject in a simulated home- use environment. All subjects will be provided with a list of tasks to complete, including providing a urine sample and operating the ACR | U.S. device on 2 mobile phones. After completing the test, the lay user will complete a post-test questionnaire. The study observer will also complete a questionnaire to collect information regarding the lay users' use of the ACR | U.S.

The device use will be compared with identified risks to determine if the percentage of failures is acceptable. Additionally, measurable usability criteria for specific, critical steps will be evaluated.

Following the usability test performed by the lay user, the subjects' urine samples will be tested by the study staff using the comparator device. These results will be considered as the "true value".

ELIGIBILITY:
Inclusion Criteria:

* Males and Females 18-80 years of age.
* Subjects diagnosed with a disease that normally represents itself with an abnormal concentration of albumin:

  * Diabetes Type I/Type II,
  * Hypertension,
  * any kidney disease,
  * other relevant conditions,
* or, subjects who are healthy or pregnant.
* Subject is familiar with the use of a smartphone.
* Subject is capable of comprehending and following instructions in English.
* Subject has facility with both hands.
* Subject is capable and willing to adhere to the study procedures.
* Subject is capable and willing to provide informed consent.

Exclusion Criteria:

* Subject has dementia.
* Subject has severe mental disorders.
* Subject cannot collect urine in a receptacle.
* Subject is visually impaired (cannot read the user manual).
* Any additional reason the study physician believes disqualifies the subject from participating in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - AccuMed research associates, Garden City, New York
  - PMG Research of Charleston, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study enrolled 250 subjects who met the inclusion criteria and performed a total of 546 tests at two U.S. clinical sites
Units Other Than Participants: Tests
Period: Overall Study
Arm/Group | ACR | U.S. Urine Analysis Test System
Started | 250; 546 Tests
Completed | 250; 546 Tests
Not Completed | 0; 0 Tests

BASELINE CHARACTERISTICS:
Arm/Group | ACR | U.S. Urine Analysis Test System
Number analyzed (Participants) | 250
Age, Continuous [Median (Standard Deviation); unit: years] | 57 (17.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139
  Male | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 241
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 52
  White | 188
  More than one race | 0
  Unknown or Not Reported | 1
Education Attainment [Count of Participants; unit: Participants]
  Less than 9 years of education | 1
  9 to 12 years of education | 27
  Over 12 years of education | 221
  Unknown | 1
Medical Background [Count of Participants; unit: Participants] — Numerous subjects participating in the study were diagnosed with more than one disease, therefore numbers add up to more than 100%.
  Participants
    Hypertension | 96
    Diabetes Type II | 45
    Kidney disease | 6
    Heart disease | 8
    Healthy | 139
    Other | 1
Concomitant Medications [Count of Participants; unit: Participants] — A list of concomitant medications taken by study participants was collected, including the medication name, dosage, route of administration, frequency and indication.
  Participants
    Use of one or more Concomitant medication(s) | 149
    No Use of Concomitant medication(s) | 101

OUTCOME MEASURES:

1. Primary Outcome: Accuracy Evaluation: The Degree of Agreement (%) of the ACR | U.S. Urine Analysis Test System as Compared to the Comparator Device
Description: The primary objective of the study is to evaluate the % exact match (percent agreement) and the % ±1 block match (percent agreement) of ACR | U.S. Urine Analysis Test System (tested by the lay user) compared to the URiSCAN Optima Urine Analyzer (the comparator device, tested by a healthcare professional user), for all reported values (blocks). Different concentrations reported by the ACR | U.S. Urine Analysis Test System were compared with results from the comparator device.
Time Frame: 2 months
Population: Each study participant was asked to perform the test twice: first, by using their preferred platform device (iOS or Android), in which usability and accuracy were evaluated; and secondly by using the other platform device, which was assessed for accuracy only. In addition, 23 spiked samples were used in order to achieve sufficient sample sizes for all analyte blocks, each sample on both platforms as well.
Measure: Count of Units; unit: Tests
Units Other Than Participants: Tests
Arm/Group | ACR | U.S. Urine Analysis Test System
Number analyzed (Participants) | 250
Number analyzed (Tests) | 546
Tests
  Overall - ACR Exact Agreement | 506
  Overall - ACR ± Block Match | 546
  Overall - Albumin Exact Agreement | 497
  Overall - Albumin ± Block Match | 546
  Overall - Creatinine Exact Agreement | 484
  Overall - Creatinine ± Block Match | 546

2. Secondary Outcome: Usability Evaluation: User Performance Analysis
Description: The usability of the ACR | U.S. Urine Analysis Test System was determined by evaluating the percentage of study subjects able to perform all required steps and successfully complete the test given only the instructions and training materials provided. In addition, each subject was asked to complete a post test questionnaire to assess the device ease of use by rating the various test steps on a scale of 1 to 5, with 5 being the easiest ("very easy") and 1 the hardest ("very hard"). This questionnaire also included understanding questions in a multiple-choice, quiz-like format, to assess the participants' understanding of essential information and key test procedures in the study.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | ACR | U.S. Urine Analysis Test System
Number analyzed (Participants) | 250
Participants
  Participants able to complete the device related tasks on 1st attempt | 250
  Overall ease of performing the test: "very easy" (5 out of 5) | 241
  Overall ease of performing the test: "easy" (4 out of 5) | 9
  Overall ease of performing the test: "normal" (3 out of 5) | 0
  Overall ease of performing the test: "hard" (2 out of 5) | 0
  Overall ease of performing the test: "very hard" (1 out of 5) | 0
  1st understanding question: participants who answered correctly | 241
  2nd understanding question: participants who answered correctly | 250
  3rd understanding question: participants who answered correctly | 240
  4th understanding question: participants who answered correctly | 249
  5th understanding question: participants who answered correctly | 250

ADVERSE EVENTS:
Time Frame: Up to 1 day for each patient. Monitoring of adverse events begun after the Informed Consent Form was signed and the first study-related procedure was performed and continued until the last study-related procedure was performed.
Description: The definitions are not differ from the clinicaltrials.gov definitions.
Arm/Group | ACR | U.S. Urine Analysis Test System
All-Cause Mortality (participants affected / at risk) | 0/250
Serious Adverse Events (participants affected / at risk) | 0/250
Other Adverse Events (participants affected / at risk) | 0/250

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT04626271/Prot_SAP_000.pdf